CLINICAL TRIAL: NCT05890248
Title: Ultrasound Guided Erector Spinae Block Versus Thoracic Para-vertebral Block Versus Quadratus Lamborum Block in Open Renal Surgeries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: mohamed A Aboelsuod, MD (Other)
Responsible Party: Sponsor-Investigator, mohamed A Aboelsuod, MD, assisstant professor, Al-Azhar University
Organization: Al-Azhar University (Other)
Other Study IDs: Mohamed A Aboelsuod
Record Dates: First submitted 2023-05-14; First posted 2023-06-06 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Erector spinea block: -ESPB Group (n=12): Received erector spinae plane block.
  Interventions: Procedure: Technique
- Thoracic Paravertebral block: TPVB Group (n=12) : Received thoracic paravertebral block.
  Interventions: Procedure: Technique
- Control group: Control Group (n=12): Received morphine (0.1 mg/kg iv) before skin incision .
- QLB group: Quadratus lamborum block n=12
  Interventions: Procedure: Technique

INTERVENTIONS:
Procedure: Technique — Paravertebral block versus Erector spinea block versus quadratus lamborum block
  Other Names: Paravertebral block versus Erector spinea block versus quadratus lamborum block
  Groups: Erector spinea block; QLB group; Thoracic Paravertebral block

SUMMARY:
Open renal surgeries are associated with substantial postoperative pain, pain relief in patients undergoing this procedure is usually provided either by thoracic epidural analgesia (EA) or by systemic analgesics. EA is a very useful option for the management of postoperative pain in patients undergoing abdominal surgeries, but the risks and contraindications linked to EA like hypotension, headache, nerve damage or infection may limit its use. Systemic analgesics in the form of opioid analgesics may give rise to side effects like nausea ,vomiting , constipation , allergy or drowsiness and often provide insufficient analgesia. Hence, other methods of postoperative pain management are desired. Sensory level target according to the incision site Flank (T9-T11) , Thoraco-abdominal (T7-T12 ) and Trans-abdominal (T6-T10). Ultrasound (US) guided erector spinae plane (ESP) block is one of the interfascial plane blocks that target the dorsal and ventral rami of the spinal nerves. Although there is no sufficient evidence for the spread of local anesthetic to the ventral rami, recent reports demonstrated effective postoperative analgesia after thoracic and lumbar surgeries affecting both the ventral and dorsal rami. Paravertebral block (PVB) is a technique where a local anesthetic is deposited into a space found on both sides of the spine, called the paravertebral space. It is a block with a dermatomal distribution of pain relief depending on the level of the spine at which the block is sited and the quantity and type of deposited local anesthetic.

PVB is effective for pain relief in the thoracic, abdominal and limb regions. primary aim was to compare postoperative opioid consumption rates at 24 h. Secondary end points were to compare pain scores and hemodynamic variables.

DETAILED DESCRIPTION:
This was randomized, controlled, single-blinded study, conducted in urology operating theatre, Al-Azhar university hospital. Forty eight patients of both sex and aged from 21-65 years in period between February 2022 to January 2023 scheduled for elective open renal surgeries under general anesthesia were enrolled in this study. The procedure was explained to the patient and informed consent was signed after his agreement then the patient was classified to one of three groups

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Adult patients of both sex, (21-65 years) with renal surgeries with ASA I , II score.

Exclusion criteria

* Patient's refusal.
* Patients with ASA (III , IV) score.
* Coagulopathy to be cancelled if ( INR>1.4 , Platelets count <100x109 )
* Infection at the injection site.
* Allergy to local anesthetics.
* Patients receiving opioids for chronic analgesic therapy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This was randomized, controlled, single-blinded study, conducted in urology operating theatre, Al-Azhar university hospital. Forty eight patients of both sex and aged from 21-65 years in period between February 2022 to September 2023 scheduled for elective open renal surgeries under general anesthesia were enrolled in this study. The procedure was explained to the patient and informed consent was signed after his agreement then the patient was classified to one of three groups
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine requirements 24 hours postoperatively | 24 hours post operative

CONTACTS AND LOCATIONS:
Locations (1):
- Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No